CLINICAL TRIAL: NCT07174570
Title: Repurposing Celecoxib to Overcome Resistance to Immunotherapy in Advanced HCC (RECON Study)
Brief Title: Celecoxib, Durvalumab and Tremelimumab for the Treatment of Patients With Advanced or Metastatic Liver Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Olumide Gbolahan, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008622; P30CA138292 (NIH); NCI-2025-06192 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP6414-24 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2025-09-11; First posted 2025-09-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Celecoxib; durvalumab; Disulfides; Immunoglobulin G; tremelimumab; Antigens; Specimen Handling; Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (celecoxib, durvalumab, tremelimumab) (Experimental): Patients receive celecoxib PO BID on days 1-28 of each cycle, durvalumab IV over 30 minutes on day 1 of each cycle and tremelimumab IV over 30 minutes on day 1 of cycle 1 only. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, CT or MRI throughout the study. Patients may undergo tissue biopsy during screening.
  Interventions: Drug: Celecoxib; Biological: Durvalumab; Biological: Tremelimumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biopsy Procedure

INTERVENTIONS:
Drug: Celecoxib — Receive by mouth (PO).
  Other Names: , Benzenesulfonamide, 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]-,; Celecoxib, celecoxib, Elyxyb, Onsenal, SC-58635, YM 177; Celebrex, Celecoxib, CELECOXIB, CELECOXIB, 169590-42-5, 4-(5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl)benzenesulfonamide
Biological: Durvalumab — Receive intravenously (IV).
  Other Names: Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer, MEDI 4736, MEDI-4736, MEDI4736; 1428935-60-7, DURVALUMAB, Durvalumab, Imfinzi, Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain)
Biological: Tremelimumab — Given intravenously (IV).
  Other Names: CP675206, Imjudo, Immunoglobulin G2, Anti-(Human CTLA-4 (Antigen)) (Human Monoclonal CP-675206 Clone 11.2.1 Heavy Chain) Disulfide with; 745013-59-6, Anti-CTLA4 Human Monoclonal Antibody CP-675,206, CP 675, CP 675206, CP-675, CP-675,206, CP-675206, CP675,
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection, Biological Sample Collection, Biospecimen Collected, Biospecimen Collection, Specimen Collection
Procedure: Computed Tomography — Undergo Computed Tomography (CT).
  Other Names: CAT, CAT Scan, Computed Axial Tomography, Computed Tomography,Computed Tomography; Computerized axial tomography, Computerized Axial Tomography (procedure), Computerized Tomography, Computerized Tomography (CT) scan, CT, CT SCAN, CT scan; Diagnostic CAT Scan Service Type, tomography
Procedure: Magnetic Resonance Imaging — Undergo Magnetic Resonance Imaging (MRI).
  Other Names: Magnetic Resonance, Magnetic Resonance Imaging; MR, MR Imaging, MRI Scan, MRI, NMR Imaging, NMRI, nuclear magnetic resonance imaging,; Nuclear Magnetic Resonance Imaging, sMRI, Structural MRI
Procedure: Biopsy Procedure — Undergo tissue biopsy.
  Other Names: Biopsy, BIOPSY, Biopsy, Biopsy, Biopsy, biopsy, Biopsy, Biopsy, Biopsy, Biopsy, Biopsy, BIOPSY_TYPE, BIOPSY_TYPE, BIOPSY_TYPE, Bx

SUMMARY:
This phase II trial tests how well the combination of celecoxib with durvalaumab and tremellimumab works in treating patients with hepatocellular cancer (liver cancer) that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). Celecoxib belongs to the family of drugs called nonsteroidal anti-inflammatory agents and is used to reduces pain. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as durvalumab and tremelimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving celecoxib with durvalaumab and tremellimumab may better treat patients with advanced or metastatic liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of the combination of celecoxib, and durvalumab+ tremelimumab in advanced hepatocellular carcinoma (HCC).

SECONDARY OBJECTIVES:

I. To evaluate the activity of the combination of celecoxib, and durvalumab+ tremelimumab in advanced HCC.

II. To evaluate the safety and feasibility of the combination of celecoxib, and durvalumab+ tremelimumab in advanced HCC.

TERTIARY/EXPLORATORY:

I. To evaluate biomarkers associated with the efficacy of the combination of celecoxib, and durvalumab+ tremelimumab in advanced HCC.

OUTLINE:

Patients receive celecoxib orally (PO) twice daily (BID) on days 1-28 of each cycle, durvalumab intravenously (IV) over 30-60 minutes on day 1 of each cycle and tremelimumab IV over 30-60 minutes on day 1 of cycle 1 only. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study. Patients may undergo tissue biopsy during screening.

After completion of study treatment, patients are followed up at 30 days, and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular cancer (HCC) planned for treatment at gastrointestinal clinics of Emory University's Winship Cancer Institute or Grady Cancer Center
* Radiologically measurable disease based on Response Evaluation Criteria in Solid Tumors version (RECIST) 1.1
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Platelet count > 100,000 cells/ ul (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Hemoglobin (Hb) > 9g/dl (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Absolute neutrophil count > 1000 cells/dl (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Albumin > 3g/dl (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Total bilirubin < 3mg/dl (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Glomerular filtration rate (GFR) > 60ml/min (based on creatine, and cystatin C estimation where applicable) (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Females of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy
* FCBP and men treated or enrolled on this protocol must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 3 months after completion of study drug administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

  * A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Completion of all previous cancer directed therapy (including, radiotherapy, liver lesion ablation, bland or chemoembolization and transarterial radioembolization therapy) ≥ 4 weeks before the start of study therapy.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class IIB or better.

  * Patients without existing cardiac disease that could raise the risk of complications who consent for the trial will proceed with trial participation
  * Patients with existing cardiac disease that could raise the risk of complications will be referred at the discretion of the investigator to a cardio-oncologist or general cardiologist for cardiac optimization prior to starting celecoxib
* Life expectancy > 12 weeks as determined by the investigator
* Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions. This includes willingness to undergo mandatory blood sample draws for evaluation of correlatives
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.

Exclusion Criteria:

* Mild to moderate liver dysfunction evidenced by Child Pugh score 7B and above
* History of arterial or venous thromboembolic events or gastrointestinal bleeding event. Subjects with portal venous thrombosis are permitted in the study if their treating oncologist does not deem it necessary to treat this with heparin products or direct acting anticoagulant (DOAC)
* Current use of warfarin, heparin products and DOACs
* Subjects with a history of (non-bleeding) peptic ulcer disease who have been on a proton pump inhibitor for less than 30 days prior to screening visit
* Patients who have had immune checkpoint inhibitors (ICI) therapy within 6 months prior to entering the study or those who have not recovered from adverse events due to liver directed therapy administered more than 4 weeks earlier (i.e., have residual toxicities > grade 2)
* Patients who are receiving any other investigational agents or an investigational device within 28 days before administration of first dose of study drugs
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in study
* Contraindication to ICI per investigator discretion
* Uncontrolled current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Significant cardiovascular disease (e.g., myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 3 months prior to start of study therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure; or uncontrolled grade ≥ 3 hypertension (diastolic blood pressure ≥ 100 mmHg or systolic blood pressure ≥ 160 mmHg) despite antihypertensive therapy
* Contraindication to non-steroidal anti-inflammatory drugs (NSAIDs): cardiac conditions that significantly raise the risk of cardiopulmonary complications, including unstable angina, uncontrolled heart failure, recent gastrointestinal (GI) bleed. Note that patients who are stable on low dose aspirin (< 325mg/day) only will be allowed on study
* Current use of other NSAIDs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-11-13 (Estimated); Study Completion 2027-11-13 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Time between the date of registration and the first date of documented progression, regardless of discontinuation of study drug, or death due to any cause, whichever occurs first, assessed up to 2 years
  PFS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median PFS will be estimated using the Brookmeyer-Crowley approach.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  ORR defined as the proportion of all subjects whose best overall response is either a complete response or partial response per Response Evaluation Criteria in Solid Tumors version 1.1 criteria. ORR will be reported as a proportion, and 95% exact binomial confidence interval will be estimated using the Clopper-Pearson method.
Incidence of Adverse Events (AE) | Up to 2 years
  Will be determined according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5. Frequencies and percentages will be used to summarize safety events.
One Treatment Cycle | During cycle 1 (cycle 1 = 28 days)
  Frequencies and percentages will be used to determine the proportion of subjects who complete one treatment cycle.
Incidence of Adverse Events Profile | Up to 2 years
  Incidence of Adverse Events (AE) profile with the combination of celecoxib, and durvalumab+ tremelumumab will be determined according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5. Frequencies and percentages will be used to summarize events.

CONTACTS AND LOCATIONS:
Overall Officials: Olumide B. Gbolahan, MBBS, MSc, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia